CLINICAL TRIAL: NCT04581044
Title: Impact of COVID-19 on Psoriasis Practice: A Cross Sectional Study
Brief Title: Impact of COVID-19 on Psoriasis Practice
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona El-Kalioby, Principal Investigator, Cairo University
Other Study IDs: KAPU2020 10
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis; Covid19
Keywords: Psoriasis; coronavirus; Sars-Cov-2
MeSH Terms: conditions — Psoriasis; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 had a major impact on dermatology practice globally with special emphasis on chronic diseases e.g. psoriasis. The main objective of this work is to investigate the effect of COVID-19 pandemic on psoriasis management.

This work is designed as a cross-sectional survey based on a questionnaire directed to Egyptian dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Dermatologists

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian Dermatologists
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Questionnaire to assess 1) Prescription pattern for Psoriasis patients during COVID-19 2) Management pattern for Psoriasis patients during COVID-19 | 2-4 weeks
Questionnaire to assess 1) Impact of COVID-19 on the course of psoriasis in patients 2) Impact of COVID-19 on the psoriasis patients behaviour | 2-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mona El-Kalioby, Cairo, Egypt